CLINICAL TRIAL: NCT03441243
Title: Evaluation of the Psychological Consequences of Complicated Childbirth
Acronym: ESPT Obst
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC18_3096_ESPT Obst
Record Dates: First submitted 2018-02-15; First posted 2018-02-22 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Parturition

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Case group:Cesarean section urgently: - 43 patients had an emergency caesarean section between 01/01/2015 and 31/12/2016.
- Case group:Hemorrhage of deliverance: - 85 patients had haemorrhage of the delivery with need for a transfusion between 01/01/2015 and 31/12/2017.
- Control group: delivery physiological low path: - A control group will consist of 128 patients who had a physiological low birth delivery over the same period.

SUMMARY:
Prospective, non-interventional, monocentric, case-control study

DETAILED DESCRIPTION:
The post-traumatic stress state affects up to 6.2% of patients at 2 months post partum.

Emergency cesarean section and rescue hemorrhage are identified risk factors for postpartum stress disorder or postpartum depression.

These complications (emergency cesarean section and hemorrhage of delivery) alter the mother-child relationship and cognitive development of the child.

The experience of an emergency Cesarean section or a haemorrhage of deliverance generates apprehension about a subsequent pregnancy. Some patients abandon a future pregnancy project for fear of reliving these experiences.

Currently, at the southern hospital, the risk factors for developing a state of post-traumatic stress are not sought by the care teams. No specific follow-up is planned for patients who have had an emergency caesarean section or hemorrhage of delivery.

The investigators wish to study the psychological consequences of emergency cesarean section and rescue haemorrhage, the risk factors for post-traumatic stress disorder after emergency cesarean section or hemorrhage of delivery, and their consequences on the mother-child relationship to better identify situations at risk of psychological trauma and provide appropriate care for patients (consultation with a postpartum psychologist).

ELIGIBILITY:
Inclusion Criteria:

* Major patients ;
* Who had hemorrhage of the transfused delivery between 01/01/2015 and 31/12/2017 or an emergency cesarean section between 01/01/2015 and 31/12/2016 or patients who gave birth physiologically paired with age, date of delivery and parity ;
* Patients who did not express their opposition to participate in the study.

Exclusion Criteria:

* Minor patients;
* Patients who do not speak and understand French;
* Major persons subject to legal protection (safeguard of justice, guardianship, guardianship), persons deprived of their liberty.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women who gave birth between 01/01/2015 and 31/12/2017
Sampling Method: Non-Probability Sample
Enrollment: 256 (Actual)
Dates: Start 2018-05-23 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-02-27 (Actual)

PRIMARY OUTCOMES:
Post-traumatic stress | Baseline
  Post traumatic stress state score according to the PCL-5 (Posttraumatic Stress Disorder Checklist-5)

SECONDARY OUTCOMES:
Tocophobia | Baseline
  Tocophobia score according to the Tocophobia Questionnaire
Peritraumatric dissociation | Baseline
  Peritraumatric dissociation score according to the PDEQ (Peritraumatric dissociative Expériences Questionnaire)
Postpartum depression | Baseline
  Postpartum depression score according to the Edingburgh Perinatal Depression Questionnaire
Mother-child relationship | Baseline
  Mother-child Relationship score according to the Parent Bonding Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Dayan, Principal Investigator — Hospital-University Psychiatry Center for Children and Adolescents
Locations (1):
- Hospital-University Psychiatry Center for Children and Adolescents, Rennes, Britanny, France